CLINICAL TRIAL: NCT01210833
Title: Using HandTutor With Traumatic Hand Injuries: Characterizing the System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MMC10k112/2010CTIL
Record Dates: First submitted 2010-08-29; First posted 2010-09-29 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Hand Injuries
Keywords: Finger Fractures; Tendon Injuries; Soft Tissue Injuries
MeSH Terms: conditions — Hand Injuries; Tendon Injuries; Soft Tissue Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy participants (Active Comparator): Healthy participants aged from 18 to 60 with no history of hand injuries recruited by convenience sampling.
  Interventions: Device: HandTutor System
- Hand Injured participants (Experimental): Participants with hand injuries aged from 18 to 60 recruited from the outpatients attending the occupational therapy clinic.
  Interventions: Device: HandTutor System

INTERVENTIONS:
Device: HandTutor System — Computerized system designed to evaluate and rehabilitate hand function. It is composed of a glove with special sensors detecting the movements of the wrist and the fingers, with a biofeedback software designed to evaluate and then to exercise the hand movements through supplying a variety of computer graphic patterns.

SUMMARY:
HandTutor is a computerized system designed to evaluate and rehabilitate hand function. It is composed of a glove with optic sensors detecting the movements of the wrist and the fingers with a biofeedback software designed to evaluate and then to exercise the hand movements through supplying a variety of computer graphic patterns.

The HandTutor has been used and tested with a stroke population, and it seems potential to be used with hand injuried population. As a first step, it is important to investigate the characteristics of the system and how it is matching the hand injuried population.

The purpose if this study is to characterize the HandTuror system and the focused objectives are:

1. To examine the test-retest reliability of the system when measuring the range of motion (ROM) of the the fingers among healthy people (control group).
2. To examine the correlation between the ROM measured by the HandTutor and the ROM measured by conventional assessment tools (goniometer).
3. To examine the ability of the system to distinguish between healthy people and hand injured people.
4. To examine the correlation between the performance in the HandTutor (in the games part), and the performance in functional activities.
5. To examine the participants feedback for using the HandTutor (degree of enjoyment).

ELIGIBILITY:
Inclusion Criteria:

* Hand Injuries causing a disfunction of one finger or more of the fingers 2nd-5th.
* Six weeks at least after the injury/surgery.
* Allowed to exercise their fingers with no contraindications according to the orthopedic surgeon instructions.
* With no open wounds.

Exclusion Criteria:

* Peripheral nerves injuries.
* Digital nerves injuries.
* Sensation problems.
* CRPS-complex regional pain syndrome.
* Cognitive impairments.
* Head trauma.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
range of movement (ROM) | up to 12 months after the injury
  Passive and active ROM measured by goniometer, passive and active ROM measured by HandTutor

SECONDARY OUTCOMES:
performance in HandTutor | up to 12 months after the injury
  The final score the participants get when exercising with the HandTutor.
daily life functioning | up to 12 months after the injury
  Measured by DASH-Disability of Arm,Shoulder and Hand Questionnaire, and by Jebsen-Taylor Hand Function Test.
motor performance skills | up to 12 months after the injury
  Measured by Purdue Pegboard Test
enjoyment | up to 12 months after the injury
  Measured by SFQ-Specific feedback questionnaire.
pain | up to 12 months after the injury
  Measured by VAS-Visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Manal A. Najjar, M.Sc. in O.T, Study Director — Clalit Health Service, Southern Clinic, Occupational Therapy Department, Naẕerat 'Illit, Israel, 04-6557444, manalaz@clalit.org.il
Locations (1):
- Clalit Health Service, Southern Clinic, Occupational Therapy Department, Naẕerat ‘Illit, Israel